CLINICAL TRIAL: NCT03930745
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Of TOL-463 Insert for Suppression Of Bacterial Vaginosis (BV) [SUBVert]
Brief Title: Suppression Of Bacterial Vaginosis (BV) [SUBVert]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0017
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2020-05-27

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial vaginosis; Candida albicans; Double-Blind; Gardnerella vaginalis; Phase II; Placebo; Randomized; Suppression; TOL-463 insert
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — TOL-463

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): TOL-463 insert administered vaginally twice a week for twelve weeks. N=125
  Interventions: Drug: TOL-463
- Arm 2 (Placebo Comparator): Matching placebo insert administered vaginally twice a week for twelve weeks. N=125
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo vaginal inserts.
  Arms: Arm 2
Drug: TOL-463 — TOL-463 is a non-azole vaginal anti-infective drug candidate designed as a dual-indication therapy for BV and VVC.
  Arms: Arm 1

SUMMARY:
A Phase II randomized, double-blind, placebo-controlled study screening approximately 600 adult females, aged 18-55, with a goal to enroll approximately 250 participants to achieve 200 evaluable participants at the test of cure (TOC) visit. The study is designed to determine the clinical efficacy of an investigational product (IP), TOL-463 Insert, in suppressing Recurrent Bacterial Vaginosis (RBV) when administered to women who have a history of RBV and have been successfully cleared of their current Bacterial Vaginosis (BV) infection administering 500 mg of oral metronidazole, twice a day for 7 days or another CDC-recommended BV treatment. Patient participation will be approximately 100 days while the study is conducted at 4 sites within the United States. The primary objective of the study is to evaluate the clinical efficacy of a twice-weekly application of TOL-463 vaginal insert in suppression of BV in women with a history of RBV following successful induction with oral metronidazole or a CDC-recommended BV treatment.

DETAILED DESCRIPTION:
This is a Phase II randomized, double-blind, placebo-controlled study screening approximately 600 adult females, aged 18-55, with a goal to enroll approximately 250 participants to achieve 200 evaluable participants at the test of cure (TOC) visit. The study is designed to determine the clinical efficacy of an investigational product (IP), TOL-463 Insert, in suppressing Recurrent Bacterial Vaginosis (RBV) when administered to women who have a history of RBV and have been successfully cleared of their current Bacterial Vaginosis (BV) infection administering 500 mg of oral metronidazole, twice a day for 7 days or another CDC-recommended BV treatment. Patient participation will be approximately 100 days while the study is conducted at 4 sites within the United States. The primary objective of the study is to evaluate the clinical efficacy of a twice-weekly application of TOL-463 vaginal insert in suppression of BV in women with a history of RBV following successful induction with oral metronidazole or a CDC-recommended BV treatment. Secondary objectives of the study are: 1) to evaluate the time to BV recurrence as defined by clinical criteria, 2) to evaluate the incidence of vaginal symptoms over study participation, 3) to evaluate acceptability of a twice-weekly application of TOL-463 vaginal insert in suppression of BV, and 4) to evaluate the safety of TOL-463 vaginal insert compared to placebo, including the incidence of secondary vulvovaginal candidiasis (VVC). The null hypothesis for the comparison is that there is no difference in cure rates between treatments, with a two-sided alternative.

ELIGIBILITY:
Inclusion Criteria:

Screening Visit(s) Inclusion Criteria:

1. Women with a current Bacterial Vaginosis (BV) infection and a history of at least two previous episodes of BV by documentation or self-report in the past year. Screening (V0) diagnosis is based on the presence of > / = 3 Amsel criteria*;

   * Homogeneous vaginal discharge; positive potassium hydroxide (KOH) whiff test; vaginal pH of > 4.5; and > / = 20% clue cells.
2. Willing and able to provide written informed consent;
3. Age 18-55 years of age at the time of V0;
4. General good health based on medical history, targeted physical examination, and pelvic examination;
5. For participants 21 years of age or older, Pap test performed within the past 3 years, with the most recent result being normal or Atypical Squamous Cells of Undetermined Significance (ASCUS) Human Papillomavirus (HPV) negative or Pap smear collected at V0*;

   *Consistent with current Pap screening guidelines, a Pap smear must be performed at V0, for women who meet the following criteria and cannot provide documentation or self-report of a normal or ASCUS HPV negative Pap smear, conducted within the prior 3 years: (a) has not had a hysterectomy or (b) has had a hysterectomy and has a history of cervical intraepithelial neoplasia grade 2 plus (CIN2plus) in the past 20 years.

   Note: If a Pap smear is conducted at V0, the results are not required prior to enrollment.
6. Have a negative urine pregnancy test at V0, if of childbearing potential;
7. Must be of non-childbearing potential* or must be using an effective method of birth control** and must be willing to continue the method through the end of Investigational Product (IP) administration;

   *Defined as post-menopausal or status post bilateral tubal ligation, or status post bilateral oophorectomy or status post hysterectomy.

   **Acceptable methods are defined as:
   1. Intrauterine Devices (IUDs) or hormonal contraceptives for at least 22 days prior to screening. Note: Intravaginal contraceptive rings (e.g., NuvaRing) are not acceptable forms of birth control for this study.
   2. Consistent use of a barrier method, including diaphragms or condoms, for at least 13 days prior to screening.
   3. Abstinence from vaginal sexual intercourse for at least 13 days prior to screening.
   4. Exclusively same-sex relationship.
   5. Monogamous relationship with vasectomized partner.
8. Willing and able to cooperate to the extent and degree required by this protocol at the discretion of the investigator;

Enrollment Visit Inclusion Criteria:

In addition to confirming all relevant Screening Visit Inclusion Criteria, women must meet all of the following criteria to be eligible for enrollment in the study.

1. Willing and able to provide Enrollment written informed consent;
2. After completion of metronidazole induction therapy or another CDC-recommended BV treatment, no clinical evidence of BV* and absence of symptoms of BV** at Visit 1, Enrollment (V1);

   * As defined by < / = 2 of 4 Amsel criteria. **Defined as absence of vaginal discharge and odor consistent with BV.
3. Must have a negative urine pregnancy test at V1, if of childbearing potential;
4. Willing to refrain from any intravaginal products/medications* other than the IP throughout the course of the trial;

   *For example: douches, antifungal or antibacterial preparations, lubricants, contraceptive creams, gels, foams, sponges, spermicides.
5. Must agree to abstain from receptive oral, anal, and vaginal sexual intercourse one hour prior to IP administration and for 24 hours after;
6. Willing to refrain from using tampons or menstrual cups for 24 hours after IP administration;
7. Must be of non-childbearing potential* OR must be using an effective method of birth control** and must be willing to continue the method through the end of IP administration; *Defined as post-menopausal or status post bilateral tubal ligation, or status post bilateral oophorectomy or status post hysterectomy.

   * Acceptable methods are defined as:

     1. IUDs or hormonal contraceptives for at least 30 days prior to using IP. Note: Intravaginal contraceptive rings (e.g., NuvaRing) are not acceptable forms of birth control for this study.
     2. Consistent use of a barrier method, including diaphragms or condoms, for at least 21 days prior to using IP.
     3. Abstinence from vaginal sexual intercourse for at least 21 days prior to using IP.
     4. Exclusively same-sex relationship.
     5. Monogamous relationship with vasectomized partner.

Exclusion Criteria:

Screening Visit(s) Exclusion Criteria:

1. Diagnosis of another vaginal or vulvar condition that may confuse interpretation of response to Investigational product (IP)*;

   * For example: erosive lichen planus, desquamative inflammatory vaginitis, or contact dermatitis involving the vulvar epithelium.
2. Concurrent Vulvovaginal Candidiasis (VVC) infection with inability to be treated with oral fluconazole;
3. Infectious cause of cervicitis (e.g., N. gonorrhoeae, C. trachomatis, or T. vaginalis) confirmed on physical examination and/or with laboratory testing*, **;

   *Women may be rescreened for eligibility following successful treatment of confounding Sexually Transmitted Infection (STI).

   **Results of Nucleic Acid amplification Test (NAAT) testing will be reviewed prior to enrollment.
4. Active genital lesions, including ulcers or vesicles consistent with herpes or warts;
5. Planned ongoing immunosuppressive therapy or systemic antibiotic treatment during the course of the study;
6. History of hypersensitivity, allergy or other contraindication(s) to metronidazole or other CDC-recommended BV treatment used to treat subject;
7. History of hypersensitivity to any TOL-463 formulation components;
8. Current or untreated cervical intraepithelial neoplasia (CIN) or cervical carcinoma;
9. Currently pregnant or nursing;
10. Any other condition that, in the opinion of the investigator, would interfere with participation in the study;
11. Previous enrollment in the study or at the investigator's discretion;

Enrollment Visit Exclusion Criteria:

In addition to confirming all Screening Visit Exclusion Criteria, women who meet any of the following criteria will not be eligible for enrollment in the study.

1. Active menses or significant vaginal bleeding as determined by the study clinician at V1*;

   *Note: women who are menstruating may be reevaluated for study enrollment within the enrollment window.
2. Use of vaginal or systemic antibiotic or antifungal since V0, other than oral metronidazole, CDC-recommended BV treatment, or oral fluconazole, as per protocol;
3. Evidence or suspicion of infectious cause of cervicitis or active genital lesion on pelvic examination at Visit 1, Enrollment (V1);
4. Concurrent VVC infection at V1 with inability to treat with oral fluconazole;
5. Use of any investigational drug within 30 days prior to V1 or planned/anticipated use during study participation.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 81 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - University of California, San Diego - Antiviral Research Center, La Jolla, California
  - Cook County Health and Hospitals System - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Magee Women's Hospital of UPMC - Reproductive Infectious Disease Research, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adult females 18-55 years of age with a history of recurrent bacterial vaginosis. Participants were recruited from United States health clinics and enrolled between 09SEP2019 and 20SEP2021
Groups:
- TOL-463 Vaginal Insert: TOL-463 Vaginal Insert administered vaginally as a single 2 gram unit dose twice a week with a minimum of a two-day duration in between doses for twelve weeks with the aid of a disposable applicator.
  TOL-463 Vaginal Insert: Non-azole vaginal anti-infective drug candidate designed as a dual-indication therapy for bacterial vaginosis (BV) and vulvovaginal candidiasis (VVC). Hydrophilic melt insert supplied in 2.0 cc/g low density polyethylene (LDPE) + polyvinyl chloride (PVC) plastic unit-dose insert molds with ten vaginal applicators.
- Placebo: Placebo administered vaginally as a single 2 gram (g) unit dose twice a week with a minimum of a two-day duration in between doses for twelve weeks with the aid of a disposable applicator.
  Placebo: Matching placebo vaginal insert supplied in 2.0 cc/g low density polyethylene (LDPE) + polyvinyl chloride (PVC) plastic unit-dose insert molds with ten vaginal applicators.
Period: Overall Study
Arm/Group | TOL-463 Vaginal Insert | Placebo
Started | 40 | 41
Completed | 24 | 25
Not Completed | 16 | 16
Not completed — Lost to Follow-up | 10 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — COVID-19 Shelter in Place Order | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- TOL-463 Vaginal Insert: TOL-463 Vaginal Insert administered vaginally as a single 2 gram unit dose twice a week with a minimum of a two-day duration in between doses for twelve weeks with the aid of a disposable applicator.
- Placebo: Placebo administered vaginally as a single 2 gram (g) unit dose twice a week with a minimum of a two-day duration in between doses for twelve weeks with the aid of a disposable applicator.
- Total: Total of all reporting groups
Arm/Group | TOL-463 Vaginal Insert | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7.3) | 34.0 (7.8) | 33.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 36 | 36 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 22 | 51
  White | 5 | 11 | 16
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81
Number of BV Occurrences in Past 12 Months Prior to Screening [Mean (Standard Deviation); unit: occurrences] | 5.3 (2.5) | 4.9 (2.7) | 5.1 (2.6)
Culture Confirmed Vulvovaginal Candidiasis (VVC) Status at Baseline [Count of Participants; unit: Participants]
  Positive | 4 | 5 | 9
  Negative | 36 | 35 | 71
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Recurrent Bacterial Vaginosis (RBV) by Visit 4, as Defined by Presence of at Least 3 Amsel Criteria
Description: Recurrent bacterial vaginosis (RBV) was defined as the presence of at least three out of the following four Amsel criteria: positive KOH whiff test, homogeneous discharge characteristic of BV, clue cells comprising at least 20% of vaginal squamous epithelial cells, and vaginal pH > 4.5. Participants who had post-baseline efficacy results but were lost to follow-up before study completion were considered "treatment failures" and counted toward the number of participants with recurrence of BV.
Time Frame: Day 1 through Day 91
Population: The modified intent-to-treat (mITT) population includes all randomized participants with negative STI results at screening and, for participants 21 years and older, either a normal or atypical squamous cells of undetermined significance (ASCUS) HPV-negative Pap test performed at screening or within the past 3 years. This analysis includes all participants in the mITT population except those with no post-baseline efficacy data available.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 31 | 33
proportion of participants | 0.581 [0.408 to 0.736] | 0.697 [0.527 to 0.826]

2. Secondary Outcome: Time to Bacterial Vaginosis (BV) Recurrence, as Defined by Presence of at Least 3 Amsel Criteria
Description: Recurrent bacterial vaginosis (RBV) was defined as the presence of at least three out of the following four Amsel criteria: positive KOH whiff test, homogeneous discharge characteristic of BV, clue cells comprising at least 20% of vaginal squamous epithelial cells, and vaginal pH > 4.5. Participants who had post-baseline efficacy results but were lost to follow-up before study completion were censored in secondary time-to-event analyses. Participants with off-study diagnosis of BV were excluded from secondary time-to-event analyses.
  The median time to BV recurrence was calculated as the first event time at which the Kaplan-Meier estimator drops to or below 0.5.
Time Frame: Day 1 through Day 91
Population: The modified intent-to-treat (mITT) population includes all randomized participants with negative STI results at screening and, for participants 21 years and older, either a normal or atypical squamous cells of undetermined significance (ASCUS) HPV-negative Pap test performed at screening or within the past 3 years. This analysis includes all participants in the mITT population, excluding those with no post-baseline efficacy data available and those diagnosed with BV off-study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 30 | 32
days | NA [42 to NA] — The median time to BV recurrence and upper limit of the confidence interval could not be estimated because fewer than 50% of participants in the TOL-463 Arm experienced on-study diagnosis of BV recurrence during the follow-up period. | 46 [16 to NA] — The upper limit of the confidence interval could not be estimated because the median estimate of time to BV recurrence was also the maximum time to recurrence in the Placebo Arm during the follow-up period.

3. Secondary Outcome: Proportion of Participants Reporting Bacterial Vaginosis (BV) Symptoms - Abnormal Vaginal Discharge
Description: The BV symptoms evaluated for efficacy at each clinic visit included abnormal vaginal discharge and vaginal odor. Both symptoms were assessed by a clinician as either consistent with BV, not consistent with BV, or absent. Only symptoms deemed consistent with BV were reported as BV symptoms.
Time Frame: Assessed at Visit 1 (Day 1), Visit 2 (Window: Days 29-35), Visit 3 (Window: Days 57-63) and Visit 4 (Window: Days 85-91).
Population: The modified intent-to-treat (mITT) population includes all randomized participants with negative STI results at screening and, for participants 21 years and older, either a normal or atypical squamous cells of undetermined significance (ASCUS) HPV-negative Pap test performed at screening or within the past 3 years. This analysis includes all participants in the mITT population with data available from the corresponding visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 40 | 41
proportion of participants
  Visit 1 | 0.025 [0.004 to 0.129] | 0.000 [0.000 to 0.086]
  Visit 2: number analyzed (Participants) | 33 | 35
  Visit 2 | 0.091 [0.031 to 0.236] | 0.114 [0.045 to 0.260]
  Visit 3: number analyzed (Participants) | 18 | 16
  Visit 3 | 0.056 [0.010 to 0.258] | 0.063 [0.011 to 0.283]
  Visit 4: number analyzed (Participants) | 14 | 10
  Visit 4 | 0.000 [0.000 to 0.215] | 0.000 [0.000 to 0.278]

4. Secondary Outcome: Proportion of Participants Reporting Bacterial Vaginosis (BV) Symptoms - Vaginal Odor
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 40 | 41
proportion of participants
  Visit 1 | 0.025 [0.004 to 0.129] | 0.024 [0.004 to 0.126]
  Visit 2: number analyzed (Participants) | 33 | 35
  Visit 2 | 0.152 [0.067 to 0.309] | 0.143 [0.063 to 0.294]
  Visit 3: number analyzed (Participants) | 18 | 16
  Visit 3 | 0.056 [0.010 to 0.258] | 0.125 [0.035 to 0.360]
  Visit 4: number analyzed (Participants) | 14 | 10
  Visit 4 | 0.000 [0.000 to 0.215] | 0.100 [0.018 to 0.404]

5. Secondary Outcome: Number of Participants Satisfied With the Study Treatment as Assessed by Satisfaction Questionnaire Responses
Description: The satisfaction questionnaire contained five questions assessing participant satisfaction with the study treatment. For questions regarding ease of use, frequency of use, and overall satisfaction, participants could respond on a scale ranging from "Extremely dissatisfied" to "Extremely satisfied." Participants who responded with "Somewhat satisfied" through "Extremely satisfied" were considered "Satisfied" with those categories. For the question regarding convenience of use, participants could respond on a scale ranging from "Extremely inconvenient" to "Extremely convenient." Participants who responded with "Somewhat convenient" through "Extremely convenient" were considered "Satisfied" with study treatment convenience. For the question of whether the participant would use the study treatment again, participants who responded with "Yes" were considered "Satisfied" with the study treatment.
Time Frame: Assessed at study completion (the visit at which the participant was diagnosed with BV, or Visit 4 for participants remaining BV suppressed). This may occur at Visit 2 (Window: Days 29-35), Visit 3 (Window: Days 57-63) or Visit 4 (Window: Days 85-91).
Population: The modified intent-to-treat (mITT) population includes all randomized participants with negative STI results at screening and, for participants 21 years and older, either a normal or atypical squamous cells of undetermined significance (ASCUS) HPV-negative Pap test performed at screening or within the past 3 years. This analysis includes all participants in the mITT population who completed the satisfaction questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 27 | 33
Participants
  Ease of use: Satisfied | 25 | 28
  Ease of use: Not Satisfied | 2 | 5
  Frequency of use: Satisfied | 25 | 33
  Frequency of use: Not Satisfied | 2 | 0
  Convenience of use: Satisfied | 26 | 29
  Convenience of use: Not Satisfied | 1 | 4
  Overall satisfaction: Satisfied | 26 | 25
  Overall satisfaction: Not Satisfied | 1 | 8
  Would use study treatment again: Satisfied | 25 | 26
  Would use study treatment again: Not Satisfied | 2 | 7

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) Considered Product-related Following Initiation of Study Treatment
Description: Safety was monitored throughout the study, including via participant reporting. Study clinicians assessed whether or not reported adverse events (AEs) were related to study treatment.
Time Frame: Day 1 through Day 91
Population: The Safety population includes all randomized participants who received at least one dose of study treatment. Participants with any evidence of dosing according to memory aid or study IP packaging return were included in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 33 | 37
Participants | 11 | 10

7. Secondary Outcome: Number of Participants With Culture Confirmed Secondary VVC Following Initiation of Study Treatment
Description: Assessment of vulvovaginal candidiasis (VVC) was performed by pelvic examination at baseline and at each follow-up visit. If clinical diagnosis of VVC was determined at any visit, then a confirmatory Candida culture was performed.
Time Frame: Day 1 through Day 91
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | TOL-463 Vaginal Insert | Placebo
Number analyzed (Participants) | 33 | 37
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Safety was monitored from Visit 1 (Day 1) through Visit 4 (Window: Days 85-91).
Description: AEs were defined according to ICH E6. Any medical condition present at the time of screening was considered baseline and was not reported as an AE. If the severity of any pre-existing medical condition increased, it was recorded as an AE. AEs were collected for all enrolled participants.
Groups:
- Placebo: Placebo administered vaginally as a single 2 gram unit dose twice a week with a minimum of a two-day duration in between doses for twelve weeks with the aid of a disposable applicator.
Arm/Group | TOL-463 Vaginal Insert | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 13/40 | 9/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOL-463 Vaginal Insert (N=40) | Placebo (N=41)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Vaginal Discharge (Reproductive system and breast disorders) | 5 (5) | 3 (3)
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 4 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03930745/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03930745/SAP_001.pdf